CLINICAL TRIAL: NCT06837688
Title: Evaluation of Xenogeneic Collagen Matrix Versus Connective Tissue Graft to Enhance Soft Tissue Profile Around Single Dental Implants in the Aesthetic Zone
Brief Title: Enhancing Soft Tissues Around Inserted Implants by Two Different Methods
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Perio-01-2025
Record Dates: First submitted 2025-02-15; First posted 2025-02-20 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Missing Teeth
Keywords: Peri-implant soft tissue augmentation; Xenogeneic collagen matrix; Connective tissue graft
MeSH Terms: conditions — Anodontia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: After screening and obtaining informed consent, patients are randomly allocated into one of the two intervention groups (CTG or XCM) in a 1:1 ratio using a permuted block randomization method with block sizes of 4 and 6. The allocation sequence, generated by an independent statistician, is secured in sequentially numbered, opaque envelopes and is revealed at the time of surgery to assign the appropriate intervention. Our study is designed as a single-blinded trial. The outcome assessors and data analysts will be blinded to treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Connective tissue graft group (Active Comparator): Patients receive soft tissue augmentation using an autogenous connective tissue graft. A full-thickness flap is elevated at the implant site, and after implant placement, a CTG is harvested from the palatal mucosa. The graft is then trimmed to the defect dimensions and positioned under the flap to augment the peri-implant soft tissue. The donor site is sutured with double-cross sutures to ensure proper healing
  Interventions: Procedure: Peri-implant soft tissue augmentation using connective tissue graft
- Xenogeneic collagen matrix group (Experimental): Patients receive soft tissue augmentation using a xenogeneic collagen matrix (Mucoderm®). After implant placement and flap elevation, the XCM, initially sized at 15 × 20 mm, is moistened in saline for 10 minutes and slightly compressed. It is then adapted to the recipient site following a superficial incision to release muscle tension and secured to the buccal mucosa with single sutures. A screw-retained provisional restoration is installed immediately after surgery to support the augmented tissue.
  Interventions: Procedure: Peri-implant soft tissue augmentation using xenogenic collagen matrix

INTERVENTIONS:
Procedure: Peri-implant soft tissue augmentation using connective tissue graft — A full-thickness flap will be elevated after a crestal and sulcular incision at the single tooth gap and adjacent teeth. A surgical guide will be fitted and adjusted if needed. A dental implant will be placed as planned digitally in an optimal 3D position. A connective tissue graft (CTG) will be harvested from the palatal mucosa using the De-epithelialized free gingival graft technique and tailored to the site dimensions. The graft will be carefully positioned under the elevated flap to augment the soft tissue. The palatal wound will be sutured with double-cross sutures.
  Arms: Connective tissue graft group
Procedure: Peri-implant soft tissue augmentation using xenogenic collagen matrix — A full-thickness flap will be elevated after a crestal and sulcular incision at the single tooth gap and adjacent teeth. A surgical guide will be fitted and adjusted if needed. A dental implant will be placed as planned digitally in an optimal 3D position. The xenogenic collagen matrix, initially measuring 15 × 20 mm, is first moistened in saline for 10 minutes and slightly compressed to adapt its thickness to the defect. After a superficial incision to release any muscle tension, the XCM is accurately positioned and secured to the buccal mucosa using single sutures.
  Arms: Xenogeneic collagen matrix group

SUMMARY:
This randomized controlled clinical trial investigates the efficacy of xenogeneic collagen matrix (XCM) versus autogenous subepithelial connective tissue graft (SCTG) in enhancing the peri-implant soft tissue profile around single dental implants in the aesthetic zone of the anterior maxilla. Thirty adult patients with a single missing tooth, adequate bone volume, and sufficient keratinized tissue will be recruited at Damascus University. Each patient will undergo a fully digital workflow for implant planning-including CBCT imaging, intraoral scanning, and CAD/CAM fabrication of a surgical guide and provisional restoration-to ensure precision in implant placement. Immediately following implant insertion, patients will be randomly allocated (1:1) to either receive a CTG harvested from the palatal mucosa using a single incision technique or an XCM (Mucoderm®, Botiss Biomaterials) that is adapted and secured to the buccal mucosa. The primary outcome is the increase in buccal soft tissue profile, measured via superimposed digital surface models at baseline, immediately postoperatively, and at 3 months. Secondary outcomes include patient-reported measures (pain, edema, aesthetic satisfaction), clinical parameters (keratinized tissue width, soft tissue height), peri-implant health assessments, and radiographic assessment. By comparing these two methods, the study aims to determine whether the less invasive XCM can offer outcomes comparable to the CTG standard while reducing donor site morbidity and overall surgical time.

DETAILED DESCRIPTION:
This clinical trial is designed to evaluate and compare the performance of two soft tissue augmentation techniques-autogenous subepithelial connective tissue graft (CTG) and xenogeneic collagen matrix (XCM, Mucoderm®)-when used concurrently with dental implant placement in the aesthetic zone of the anterior maxilla. The rationale for this study stems from the clinical challenge of achieving optimal soft tissue esthetics and function following tooth loss. While CTG has long been considered the gold standard for increasing peri-implant soft tissue thickness, it requires a secondary surgical site, which may lead to donor site morbidity, limited tissue availability, and increased surgical time. In contrast, XCM offers a promising alternative that is biocompatible, readily available, and less invasive.

Patients aged 18 years or older with a single missing tooth in the aesthetic zone, adequate bucco-palatal bone (≥6 mm), and at least 5 mm of keratinized tissue width will be considered eligible for the study. The enrollment process begins with a thorough screening process involving clinical and radiographic examinations, including a low-dose, small-field CBCT scan and an intraoral scan. These imaging modalities allow for accurate digital implant planning using specialized software, ensuring optimal implant positioning. The digital data will be used to fabricate a stereolithographic surgical guide and design a custom CAD/CAM screw-retained provisional restoration.

Following successful screening and informed consent, the surgical phase commences. Under local anesthesia, a full-thickness flap is elevated at the implant site. Guided by the digital plan, a dental implant is precisely positioned using the surgical guide. At this point, participants are allocated to one of two intervention groups based on a strict randomization protocol.

In the CTG group, a connective tissue graft is harvested from the palatal mucosa using the de- epithelialized free gingival graft technique. The harvested graft is then trimmed to match the dimensions of the recipient site and carefully positioned under the elevated flap to augment the soft tissue. The donor site is sutured using gelatin matrix to ensure proper healing. This technique, while effective, is associated with postoperative discomfort and additional surgical time due to the need for a second operative site.

Conversely, in the XCM group, soft tissue augmentation is achieved using a xenogeneic collagen matrix (Mucoderm®). The graft, initially measuring 15 × 20 mm, is first moistened in saline for 10 minutes and slightly compressed to adapt its thickness to the defect. After a superficial incision to release any muscle tension, the XCM is accurately positioned and secured to the buccal mucosa using single sutures. Following soft tissue augmentation, a screw-retained provisional restoration is attached immediately, contributing to both function and esthetics during the healing phase.

The primary outcome of the study is the increase in the buccal soft tissue profile, quantitatively assessed using intraoral scans to generate digital surface models at three critical time points: preoperatively (T0), immediately after surgery (T1), and 3 months postoperatively (T2). Secondary outcomes include clinical assessments-such as probing depth, plaque index, bleeding on probing, keratinized tissue width, graft dimensions, wound closure, surgery time, and complications-as well as radiographic evaluation of marginal bone loss. In addition, patient-reported outcome measures (PROMs), including postoperative pain, swelling, aesthetic satisfaction, and willingness to undergo the same treatment again, will be recorded using validated visual analogue and Likert scales. Aesthetic outcomes, including mid-facial recession, Pink aesthetic score, and mucosal scarring index, will also be documented.

The data will be analyzed on an intention-to-treat basis by an independent statistician. Statistical comparisons between the two groups will help determine whether the xenogeneic collagen matrix offers comparable or superior results to the autogenous connective tissue graft regarding soft tissue volume augmentation, esthetic outcomes, and patient satisfaction. Ethical approval has been obtained from the University of Damascus, and the trial follows the CONSORT guidelines. The results will be disseminated through peer-reviewed publications and presentations at professional conferences, contributing valuable evidence to the field of implant dentistry.

Overall, this study is expected to provide insight into whether XCM can serve as a reliable, less invasive alternative to CTG, thereby potentially enhancing patient outcomes and reducing the complications associated with donor site morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older.
* Good oral hygiene, defined as full-mouth plaque score ≤25%.
* Having a single missing tooth in the aesthetic zone of the maxilla.
* Tooth extraction occurred at least 3 months prior to enrolment.
* Having adequate bone volume for implant placement (bucco-palatal bone dimension of at least 6 mm).
* Having at least 5 mm of keratinized tissue width at the implant site.

Exclusion Criteria:

* Systemic diseases.
* Smoking.
* Periodontal disease.
* Untreated caries lesions.
* Need for horizontal bone augmentation at the time of implant placement.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Increase in Buccal Soft Tissue Profile (BSP) | T0: Preoperative baseline. T1: Immediately after surgery. T2: 3 months postoperatively
  he BSP is defined as the volumetric change in the buccal soft tissue at the dental implant site. This outcome reflects both the thickness and contour improvements following soft tissue augmentation. Intraoral scans will be taken at three critical time points: preoperatively (T0), immediately postoperatively (T1), and 3 months postoperatively (T2). Digital surface models will be generated from these scans using specialized analysis software. The increase in BSP will be quantified as the difference in soft tissue volume (or thickness, depending on the analysis protocol) between the baseline (T0) and the 3-month follow-up (T2). Graft shrinkage will be measured between the scans immediately postoperatively (T1) and the 3-month follow-up (T2). his is a continuous variable measured in cubic millimeters (mm³) if volumetric data is used, or in millimeters (mm) if linear thickness is the chosen metric.

SECONDARY OUTCOMES:
Probing Depth (PD) | Baseline (Preoperative), 3 months, and 6 months postoperatively
  * Definition: The distance from the gingival margin to the bottom of the peri-implant pocket measured around the implant.
  * Measurement: Using a UNC-15 periodontal probe at six sites around the implant.
  * Type: Continuous variable (measured in millimeters).
Plaque Index (PI) | Baseline (Preoperative), 3 months, and 6 months postoperatively.
  * Definition: An ordinal score representing the level of plaque accumulation around the implant.
  * Measurement: Using a standardized modified plaque index (mPI).
  * Type: Ordinal variable.
Bleeding on Probing (BOP) | Baseline (Preoperative), 3 months, and 6 months postoperatively
  * Definition: The presence or absence of bleeding upon gentle probing, indicating inflammation.
  * Measurement: Using a standardized modified bleeding index (mBI).
  * Type: Binary at each site, then aggregated.
Graft Dimensions | Recorded intraoperatively.
  * Definition: The length, width, and thickness of the graft as applied.
  * Measurement: Recorded intraoperatively using a UNC-15 periodontal probe.
  * Type: Continuous variables (in millimeters).
Wound Closure | Recorded intraoperatively.
  * Definition: Wound closure is evaluated qualitatively (complete vs. incomplete).
  * Measurement: Wound closure is documented by the surgeon.
  * Type: Wound closure is categorical.
Surgery Time | immediately following surgery
  * Definition: Surgery time is the duration from the initial incision to the final suture placement.
  * Measurement: Surgery time is measured with a stopwatch.
  * Type: Surgery time is a continuous variable (in minutes).
Complications | From intervention to the end of follow-up period at 6 months.
  * Definition: Any adverse events such as infection, dehiscence, graft or implant loss.
  * Measurement: Documented by the surgical team and followed up clinically.
  * Type: Categorical (present/absent, with descriptive details).
Radiographic Evaluation of Marginal Bone Loss | Baseline (immediately postoperative), and 6 months postoperatively.
  * Definition: The change in bone level around the implant measured from the implant shoulder to the first bone-to-implant contact.
  * Measurement: Using CBCT images.
  * Type: Continuous variable (in millimeters).
Postoperative Pain and Swelling | One week postoperatively.
  * Definition: Patient's subjective rating of pain and swelling after surgery.
  * Measurement: Using a visual analogue scale (VAS) ranging from 0 (no pain/swelling) to 10 (worst possible pain/swelling).
  * Type: Ordinal variable.
Aesthetic Satisfaction | 3 months postoperatively.
  * Definition: Patient's satisfaction with the aesthetic outcome of the implant restoration and surrounding soft tissue.
  * Measurement: Using a Likert scale (1-5, where 1 is very dissatisfied and 5 is very satisfied).
  * Type: Ordinal variable.
Willingness to Undergo the Same Treatment Again | 3 months postoperatively.
  * Definition: Patient's acceptance and perceived comfort of the treatment procedure.
  * Measurement: Assessed via a Likert scale (1-5, from not willing to very willing).
  * Type: Ordinal variable.
Mid-Facial Recession | 3 and 6 months postoperatively.
  * Definition: The vertical distance from the incisal edge of the implant-supported crown to the level of the buccal mucosal margin.
  * Measurement: Using a periodontal probe.
  * Type: Continuous variable (in millimeters).
Pink Aesthetic Score (PES) | 3 and 6 months postoperatively.
  * Definition: A composite score evaluating the harmony of the peri-implant soft tissue with adjacent teeth, based on criteria such as mesial/distal papilla, tissue level, contour, and color.
  * Measurement: Using a standardized scoring system (0-14 scale).
  * Type: Ordinal variable.
Mucosal Scarring Index (MSI) | 3 and 6 months postoperatively.
  * Definition: A measure of the presence and severity of scar formation at the graft site, based on criteria like color, contour, texture, and vascularity.
  * Measurement: Assessed using a categorical scoring system.
  * Type: Categorical variable.

CONTACTS AND LOCATIONS:
Overall Officials: Suleiman Dayoub, DDS MSc PhD, Study Director — Damarcus University; Ali Omair, DDS, Principal Investigator — Damarcus University
Locations (1):
- Damascus University, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tommasato G, Del Fabbro M, Oliva N, Khijmatgar S, Grusovin MG, Sculean A, Canullo L. Autogenous graft versus collagen matrices for peri-implant soft tissue augmentation. A systematic review and network meta-analysis. Clin Oral Investig. 2024 May 5;28(5):300. doi: 10.1007/s00784-024-05684-5. PMID 38704784
- [Background] Dadlani S, Joseph B, Anil S. Efficacy of Xenogeneic Collagen Matrices in Augmenting Peri-Implant Soft Tissue: A Systematic Review and Meta-Analysis. Clin Exp Dent Res. 2024 Aug;10(4):e937. doi: 10.1002/cre2.937. PMID 39104130
- [Background] Hamdy A, Ibrahim SSA, Ghalwash D, Adel-Khattab D. Volumetric assessment of volume stable collagen matrix in maxillary single implant site development: A randomized controlled clinical trial. Clin Implant Dent Relat Res. 2024 Oct;26(5):930-941. doi: 10.1111/cid.13353. Epub 2024 Jun 27. PMID 38938060
- [Background] Surdiacourt L, Christiaens V, De Bruyckere T, De Buyser S, Eghbali A, Vervaeke S, Younes F, Cosyn J. A multi-centre randomized controlled trial comparing connective tissue graft with collagen matrix to increase soft tissue thickness at the buccal aspect of single implants: 3-Year results. J Clin Periodontol. 2025 Jan;52(1):92-101. doi: 10.1111/jcpe.13975. Epub 2024 Mar 14. PMID 38485651
- [Background] Eeckhout C, Vuylsteke F, Seyssens L, Christiaens V, De Bruyckere T, Eghbali A, Vervaeke S, Younes F, Cosyn J. A Multi-Centre Randomized Controlled Trial Comparing Connective Tissue Graft with Collagen Matrix to Increase Buccal Soft Tissue Thickness: A Cone-Beam CT Analysis. J Clin Med. 2023 Apr 19;12(8):2977. doi: 10.3390/jcm12082977. PMID 37109311
- [Background] Cosyn J, Eeckhout C, Christiaens V, Eghbali A, Vervaeke S, Younes F, De Bruyckere T. A multi-centre randomized controlled trial comparing connective tissue graft with collagen matrix to increase soft tissue thickness at the buccal aspect of single implants: 3-month results. J Clin Periodontol. 2021 Dec;48(12):1502-1515. doi: 10.1111/jcpe.13560. Epub 2021 Oct 12. PMID 34605057